CLINICAL TRIAL: NCT01684904
Title: A Phase II Trial of Proton Chemotherapy (PCT) for Resectable Esophageal or Esophagogastric Junction Cancer
Brief Title: Proton Therapy for Esophageal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5120054
Record Dates: First submitted 2012-09-07; First posted 2012-09-13 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Esophagus Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Proton radiation (Experimental): Proton radiation
  Interventions: Radiation: Proton radiation

INTERVENTIONS:
Radiation: Proton radiation

SUMMARY:
The goal of this phase II study is to investigate the feasibility, toxicity and efficacy of a regimen incorporating a proven systemic regimen, carboplatin /paclitaxel, with conformal proton modality, followed by definitive surgery. In most combined-modality trials to date, chemotherapy regimens have included cisplatin, usually in conjunction with 5-fluorouracil.

In designing the regimen, the investigators attempt to improve on the standard cisplatin/5-fluorouracil regimen in several ways. First, full-dose paclitaxel is added to the regimen. This agent has activity against advanced esophageal cancer and is also a potent radiosensitizer. Second, the substitution of carboplatin for cisplatin has resulted in reduced toxicity of various combination regimens similar to that used by CROSS trial and allows for easier administration in the outpatient setting.4 Third, for localized esophageal cancer, dose distribution patterns achievable with proton beam could potentially offer important clinical advantages relative to those achievable with x-rays (photons).19 Based on this, the investigators believe that this study should be conducted with the radiation modality that offers the best dosimetry achievable at our institution.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed primary squamous cell or adenocarcinoma of the esophagus that involves the mid, distal or esophagogastric junction. The cancer may involve the stomach up to 5 cm.
* Endoscopy with biopsy
* Stage T1N102, T2-3N0-2 according to the American Joint Committee on Cancer (AJCC) 7th edition staging, based upon the following minimum diagnostic work-up:

History/physical examination with documentation of patient's weight within 30 days of registration

Chest/Abdominal/Pelvic contrast CT within 56 days of registration

Whole body PET/CT within 56 days of registration

Endoscopic ultrasound

Patients may have regional adenopathy including para-esophageal, gastric, gastroheptaic and celiac nodes. If celiac adenopathy present, it must be ≤ 2cm.

Patients with tumors at the level of the carina or above should undergo bronchoscopy to exclude fistula

Pulmonary function test (including routine spirometry and DLCO) within 60 days prior to registration

Serum creatinine ≤ 2 x the upper limit of normal within 4 weeks of registration

Na, K, BUN, Glucose within 4 weeks prior to registration

CBC/differential within 4 weeks prior to registration with adequate bone marrow function, defined as follows:

* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
* Platelets ≥ 100,000 cell/mm3
* Hemoglobin ≥ 8.0 g/dl (Note: the use of transfusion or other intervention to achieve Hgb ≥ 8.0 is acceptable.)

Adequate liver function, defined as total bilirubin ≤ 1.5 x upper limit of normal, AST ≤ 3 x the upper limit of normal within 4 weeks of registration

Age ≥ 18

Zubrod performance status 0-2 within 4 weeks of registration

Surgical consultation to confirm that patient will be able to undergo curative resection after completion of PCT prior to registration

For women of childbearing potential, a negative serum pregnancy test within 14 days prior to registration

Women of childbearing potential and male participants must practice adequate contraception while on study

Patient must sign study specific informed consent prior to study entry

Exclusion Criteria:

Patients with cervical esophageal carcinoma

Patients with T1N0 disease and T4 disease

Prior radiation for esophageal cancer or prior chest radiotherapy

Prior chemotherapy for esophageal cancer

Evidence of tracheoesophageal fistula or invasion into the trachea or major bronchi

Prior invasive malignancy (except non-melanomatous skin cancer), unless disease free for a minimum of 2 years ( e.g. carcinoma in situ of breast, oral cavity, or cervix are permissible)

Prior radiotherapy that would results in overlap of radiation fields

Medical contraindications to esophagectomy

Prior allergic reaction to paclitaxel or carboplatin

Severe, active co-morbidity that may impact survival

Pregnancy, nursing women, or women of child bearing potential, and men who are sexually active and not willing/able to use medically acceptable forms of contraception

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2013-02-20 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
To assess overall survival of patients treated with proton-chemotherapy (PCT) followed by surgery in patients with resectable primary esophageal or esophagogastric cancer | The major analysis for reporting the initial results of treatment will be undertaken when each patient has been potentially followed for a minimum of 3 months

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | The major analysis for reporting the initial results of treatment will be undertaken when each patient has been potentially followed for a minimum of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary Yang, MD, Principal Investigator — gyang@llu.edu
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No